CLINICAL TRIAL: NCT00226018
Title: Performance of Acceleromyography With and Without Preload During Neuromuscular Blockade
Brief Title: Performance of Acceleromyography With and Without Preload
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMG01
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Acceleromyography with Hand Adapter on dominant arm
  Interventions: Device: Hand Adapter (Organon, Oss, the Netherlands)
- 2 (Active Comparator): Acceleromyography with Hand Adapter on non-dominant arm
  Interventions: Device: Hand Adapter (Organon, Oss, the Netherlands)
- 3 (Placebo Comparator): Acceleromyography without Hand Adapter on dominant arm
  Interventions: Device: Placebo
- 4 (Placebo Comparator): Acceleromygraphy without Hand Adapter on non-dominant arm
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Hand Adapter (Organon, Oss, the Netherlands) — Randomization of acceleromyography with or without Hand Adapter to dominant or non-dominant arm. Contralateral neuromuscular transmission is measured with mechanomyography (The gold standard of neuromuscular monitoring)
  Arms: 1; 2
Device: Placebo — placebo
  Arms: 3; 4

SUMMARY:
The purpose of this study is to examine the precision, bias and limits of agreement when monitoring the neuromuscular block with acceleromyography with and without preload and compare the method to the gold standard, mechanomyography.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* General anesthesia > 1 hour
* Surgery under supine position with possibility of monitoring the neuromuscular block in both arms (thumbs)
* Written informed content

Exclusion Criteria:

* Neuromuscular disorders, hepatic and renal dysfunction
* Medication expected to interfere with the neuromuscular blocking agent
* Allergy to any medication used during anesthesia
* Body weight less or exceeding 20% of the ideal body weight
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-03; Study Completion 2006-10

PRIMARY OUTCOMES:
The precision of acceleromyography with and without preload during recovery

SECONDARY OUTCOMES:
Bias and limits of agreement for acceleromyography (AMG) with and without preload compared to mechanomyography (MMG) during recovery
All the following outcomes obtained with AMG with and without preload are compared to MMG. Furthermore the responses are compared when the AMG-values are "normalized":
Bias og limits of agreement between control TOF
Onset time
Time to reappearance of T1, T2, T3 and T4
Twitch height of T1 at reappearance of T1, T2, T3 and T4
Time to T1=25%
Interval 25-75%
Time to TOF-ratio = 0.9 and 1.0
Time to final T1
Time to final TOF ratio

CONTACTS AND LOCATIONS:
Overall Officials: Casper C Kjaer, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Dep. of anesthesia, HOC, Rigshospitalet, Copenhagen, Copenhagen Ø, Denmark